CLINICAL TRIAL: NCT05119517
Title: Can the Osteopathic Pedal Pump Reduce Lymphedema in the Lower Extremities in the Elderly? A Mentorship Project.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2020-72
Record Dates: First submitted 2021-10-29; First posted 2021-11-15 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Lymphedema, Lower Limb
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic manipulative medicine pedal pump (Experimental)
  Interventions: Other: Osteopathic manipulative medicine pedal pump

INTERVENTIONS:
Other: Osteopathic manipulative medicine pedal pump — In this 7 minute intervention, the patient receives 2 minutes of myofascial release of the thoracic inlet and then 5 minutes of the pedal pump technique

SUMMARY:
Chronic lymphedema is defined as swelling or edema (excess fluid in the interstitial space) that does not fully resolve overnight by elevating the limb or body part to the level of the heart. Chronic lymphedema is a major clinical problem that is difficult to treat. Osteopathic Pedal Pump is a simple manipulation technique anecdotally thought to reduce leg edema and chronic lymphedema. However, the clinical evidence is only anecdotal and no clinical trials have ever been conducted to test this observation. The purpose of the research is to measure the effectiveness of the Osteopathic Pedal Pump technique for treating lymphedema by measuring before and after treatment limb volumes. The second purpose of this project is to mentor osteopathic medical students in clinical research. There is also a great need to mentor Osteopathic Medical Students because relatively few pursue careers involving clinical research and the benefits osteopathic manipulative treatment remain under investigated.

ELIGIBILITY:
Inclusion Criteria:

* For phase one subjects must be age 18 or older, be a medical students at Rowan University School of Osteopathic Medicine and not have leg edema which does not resolve with overnight limb elevation. For phase two subjects must be patients at the NJISA in Stratford, NJ age 55 and over and have lower limb lymphedema. Lymphedema is defined as edema that does not resolve with overnight elevation of the lower limb.

Exclusion Criteria:

* Exclusion criteria is the same for both phases. Because the measurements involve placing the lower limb into water subjects with an open wound, sore or cellulitis in the lower limbs will be excluded to ensure good hygiene. Because lymphatic pumping can cause a redistribution of volume in the body, subjects with decompensated heart failure, acute asthma, COPD exacerbation, or active cancer will be excluded. For obvious reasons, those with a non-healed or healing bone fractures will be excluded. Due to potential problems with informed consent those with a diagnosis of dementia on the chart problem list will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Change in lower limb volume | Baseline and 1-minute after receiving pedal pump protocol
  Patient's lower limb volume measured via volumetric edema gauge

CONTACTS AND LOCATIONS:
Overall Officials: Donald Noll, DO, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States